CLINICAL TRIAL: NCT01796600
Title: Assessment of Distal Limbs Fractures With Cone-Beam CT Newtom 5G
Acronym: FRADICOBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2012.710
Record Dates: First submitted 2012-10-30; First posted 2013-02-22 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Distal Limbs Bones Fractures
Keywords: distal limbs fracture, acute trauma, imaging, cone beam computed tomography,

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Conventional and a cone-beam scanner 5G (Experimental): The patients will have a conventional scanner, a reference examination, and a cone-beam scanner Newtom 5G just after the conventional scanner
  Interventions: Device: The patients will have a conventional scanner, a reference examination, and a cone-beam scanner Newtom 5G just after the conventional scanner

INTERVENTIONS:
Device: The patients will have a conventional scanner, a reference examination, and a cone-beam scanner Newtom 5G just after the conventional scanner

SUMMARY:
ConeBeam scanner (CBCT) is a widely technique used for dental and maxillofacial imaging. Patients can be set up in a sitting or a laying position in the, Newtom 5G CBCT allowing for an analysis of the distal appendicular skeleton. The investigators' hypothesis is that the cone-beam scanner could detect and characterize fractures of the extremities similarly to a multidetector CT (MDCT). 150 patients over 18 years requiring a CT scan for a suspected distal limb fracture or a preoperative assessment will be enrolled. The primary endpointis based on the ability of cone-beam scanner to properly characterize the type of fracture using a classification derived from Maurice E. Müller (AO) classification. Secondary endpoints will concern the depiction of the fracture, the assessment of the soft tissues near the fracture, quality of images, inter and intra-operator reproducibility and tolerance of the patient for the examination. Patients will have a MDCT considered as the reference exam, then a CBCT. Exams will be anonymized and read twice by two trained radiologists with 3-6 week intervals. The inter-observer agreement for the diagnosis of fracture type between the two techniques will be evaluated by a kappa coefficient. The evaluation of diagnostic performance will be achieved by studying the sensitivity, specificity, negative predictive value and positive predictive value, and its likelihood ratio. Kappa test will be performed to evaluate the consistency of the characterization of the fracture and the evaluation of soft tissue near the fracture. A Student t test will be performed for paired data if distributions are normal, a Wilcoxon test if not. To assess patient's tolerance, the percentages of (painful, not painful) will be calculated for each technique and will be compared using the Chi2 test (or Fisher's exact test if the chi can not apply).

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years old or above, weight ≤ 160 Kg
* Patient require MDCT for a suspected distal limb fracture or a preoperative assessment
* French spoken an read
* Free and informed consent signed
* Being affiliated to a French social security system or similar.

Exclusion Criteria:

* Patients already included in the study for a previous fracture
* Patient with severe pain and reduced spontaneous mobility that could prevent proper positioning for the cone-beam
* Lack of effective contraception (risk of pregnancy) or pregnancy proven data on interrogations
* Patient on protection of the court, under supervision or trusteeship
* Inability to express a consent
* Patients already enrolled in a study with a conflict of interest with this study.
* The presence of osteosynthesis materiel or capital may interfere with image quality. A sample of 3 to 5 patients may be included at the beginning of the study to test the image quality in presence of material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Characterization of the type of fracture using a classification derived from Maurice E. Müller (AO) classification | From the day of the trauma for acute injuries to the first weeks when an occult fracture is suspected

SECONDARY OUTCOMES:
Assessment of soft tissues peripheral to the fracture | Baseline only, the day the scanner is performed.
  Articular fluid, hematoma, tendinous or ligamentous lesions
Image quality (for CBCT and MDCT) | Baseline only, the day the scanner is performed
  0 - Insufficient, 1 - Poor, 2 - Average, 3 - Good, 4 - Excellent
Tolerability and duration of the exam (for CBCT and MDCT) | Baseline only, the day the scanner is performed
  Perfect, tolerable, hardly tolerable, intolerable
Duration of the exam (for CBCT and MDCT) | Baseline only, the day the scanner is performed
  Perfect, tolerable, hardly tolerable, intolerable
Inter-intra-observer reproducibility | Bseline only, the scanner is performed.
  2 readings for each operator, with consensus reading for disagreements

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste PIALAT, MD,PHD, Principal Investigator — Hospices Civils de Lyon- Hôpital Edouard Herriot
Locations (1):
- Hospices Civils de Lyon- hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Background] Dubreuil T, Mouly J, Ltaief-Boudrigua A, Martinon A, Tilhet-Coartet S, Tazarourte K, Pialat JB. Comparison of Cone-Beam Computed Tomography and Multislice Computed Tomography in the Assessment of Extremity Fractures. J Comput Assist Tomogr. 2019 May/Jun;43(3):372-378. doi: 10.1097/RCT.0000000000000843. PMID 30762657